CLINICAL TRIAL: NCT02872792
Title: Early Mobilisation in Intensive Care Unit : Interest of Cyclo-ergometry in Patients With Septic Chock
Acronym: MUEVELO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/211/HP
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Sepsis
Keywords: cycloergometer
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early mobilisation with cyclo ergometer (Experimental): Early mobilisation with cyclo ergometer in addition of Standard physiotherapy during sepsis for patient with sepsis in ICU
  Interventions: Device: Early mobilisation with cyclo ergometer; Other: Standard physiotherapy
- Standard physiotherapy (Active Comparator): Standard physiotherapy during sepsis for patient with sepsis in ICU
  Interventions: Other: Standard physiotherapy

INTERVENTIONS:
Device: Early mobilisation with cyclo ergometer — Early mobilisation with cyclo ergometer is done daily during hospitalization for sepsis in an Intensive Care Unit
  Arms: Early mobilisation with cyclo ergometer
Other: Standard physiotherapy — Standard physiotherapy included passive and active manual mobilization, sitting on bed, sitting in chair, walking

SUMMARY:
Cycloergometer is a validated method for different care. This kind of device allow passive and active care for patient. The interest of cycloergometer for patient hospitalized in Intensive Care Unit for Sepsis has never been demonstrated.

The main objective of this study is to determine the impact of early mobilization by cyclo-ergometer in association with standard physiotherapy, on the ICU length in patients with septic shock

The secondary objectives of this study are to assess the impact of early mobilization by cyclo-ergometer in association with standard physiotherapy on:

1. the duration between hemodynamic stability* and the removal of sedation
2. the duration between the removal of sedation and ICU discharge
3. the mechanical ventilation duration (invasive and noninvasive)

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in ICU
* Septic shock diagnosed more than 24 hours before inclusion
* Patient hemodynamically stable, before the 72th hour following the diagnosis of septic shock
* Mechanical ventilation by tracheal intubation
* Patient sedated with a RASS score inferior or equal to -2
* Age ≥ 18 years
* BMI ≤ 40 kg / m²
* Informed patient having signed the consent
* Effective contraception in women of childbearing age (pregnancy test by B-HCG will be done; for menopausal women, a diagnosis of confirmation must be obtained).

Exclusion Criteria:

* BMI> 40kg / m²
* Patient reduced by one or two lower limbs
* Rheumatological pathology, trauma or surgery of the lower limbs, pelvis or spine resulting of any limitations of the range of motions or strict immobilization
* Brain-injured patient and / or medulla injured
* Hemodialysis continues with a femoral catheter without possibility of changing the catheter location
* Moribund patient, Stop or Limitation of Active Therapeutics' decision
* Contraindications to standard physical therapy or the cyclo-ergometer
* Untreated orthopedics: deep vein thrombosis of the member concerned
* Dermatological: severe lesions or complex dressings in the sector concerned
* Patient with ExtraCorporeal Membrane Oxygenation (ECMO)
* Pregnant or breastfeeding women
* Patient participating in another trial with the same main objective

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Number of days between hemodynamic stability and ICU discharge | approximately 1 month
  Number of days between hemodynamic stability (after beginning of hospitalization for sepsis) and ICU discharge

SECONDARY OUTCOMES:
Number of days between hemodynamic stability and the removal of sedation | From 3 to 10 days
  Number of days between hemodynamic stability (after beginning of hospitalization for sepsis) and the removal of sedation
Number of days under mechanical ventilation (invasive and noninvasive) during hospitalization in ICU | From 3 to 10 days
  Number of days under mechanical ventilation (invasive and noninvasive, (after beginning of hospitalization for sepsis) ) during hospitalization in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Gaétan BEDUNEAU, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No